CLINICAL TRIAL: NCT06449950
Title: The Evaluation of the Effects of Verbal and Video-Based Instructions on the Improvement of Oral Hygiene Status in Children: A Randomized Clinical Trial
Brief Title: The Effects of Different Oral Hygiene Instructions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Akif Demirel, Associate Professor, Ankara University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 11/02
Record Dates: First submitted 2024-06-04; First posted 2024-06-10 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Oral Hygiene Education; Oral Hygiene Education Methods
Keywords: Oral health education; Oral hygiene; Pediatric dental patients; Toothbrushing

STUDY DESIGN:
Intervention Model Description: For each age group (6-9 and 10-12) participants were randomly assigned to verbal and video-based oral hygiene instruction groups.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor -performing the final examination- carried out the final OHI-S index scoring blindly without knowing which Oral Hygiene Instruction group (verbal and video-based) the participants were in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Verbal Oral Hygiene Instruction Group (Experimental): Verbal oral hygiene instructions were given to the pediatric patients by the instructor using the Bass brushing technique without any training model or visual aids, only with the verbal instructions.
  Interventions: Behavioral: Behavioral: Verbal Oral Hygiene Instructions
- Video-Based Oral Hygiene Instruction Group (Experimental): The video-based oral hygiene instructions to be delivered to the paediatric dental participants were given by watching a pre-prepared video tape on a tooth and jaw model, using the instructions specified in the verbal education.
  Interventions: Behavioral: Behavioral: Video-Based Oral Hygiene Instructions

INTERVENTIONS:
Behavioral: Behavioral: Verbal Oral Hygiene Instructions — OHI-S index scores of patients who received verbal oral hygiene education were measured at baseline and final (in post-education).
  Arms: Verbal Oral Hygiene Instruction Group
Behavioral: Behavioral: Video-Based Oral Hygiene Instructions — OHI-S index scores of patients who received video-based oral hygiene education were measured at baseline and final (in post-education).
  Arms: Video-Based Oral Hygiene Instruction Group

SUMMARY:
The aim of this study is to evaluate the effects of verbal and video-based oral hygiene instructions on the oral health parameters in patients of different age groups. 202 patients in 6-9 and 10-12 aged (n=101 and n=101, respectively) were included in the study protocol. Before oral hygiene instructions, baseline oral g of all patients were determined using Simplified Oral Hygiene Index (OHI-S). Within each age group, approximately half of the participants randomly assigned to verbal (n=50 for 6-9 ages, n=51 for 10-12 ages) and video-based OHI (n=51 for 6-9 ages, n=50 for 10-12 ages). Patients were re-called for after 30 days and final OHI-S scores were recorded.

DETAILED DESCRIPTION:
In pediatric dentistry, preventive dental approaches are essential in providing sustainable oral health of children. Despite all the preventive applications, dental caries is still an important public health problem affecting preschool and school children. Oral hygiene education has an important role on the dental health services. This aims to increase awareness of oral health, provide information about it and encourage individuals to maintain oral health. Based on, the current study aims to evaluate the effects of verbal and video-based oral hygiene instructions on the oral health parameters in patients of different age groups. 202 patients in 6-9 and 10-12 aged (n=101 and n=101, respectively) were included in the study protocol. Before oral hygiene instructions, baseline oral g of all patients were determined using Simplified Oral Hygiene Index (OHI-S). Within each age group, approximately half of the participants randomly assigned to verbal (n=50 for 6-9 ages, n=51 for 10-12 ages) and video-based OHI (n=51 for 6-9 ages, n=50 for 10-12 ages). Patients were re-called for after 30 days and final OHI-S scores were recorded. Data were analysed with Shapiro-Wilk, Mann-Whitney U and Wilcoxon Signed Rank tests. Statistical significance level was considered as 5%.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 6-9 years or 10-12 years
* Children who were medically free of chronic/systemic conditions
* Patients without physical or mental disabilities or syndromes
* Patients without motor dysfunction diseases
* Patients whose permanent central incisor and permanent first molar teeth had erupted and had not been extracted for any reason

Exclusion Criteria:

* Children aged <6 or >12 years
* Children with chronic/systemic conditions
* Patients with physical or mental disabilities or syndromes
* Patients with motor dysfunction diseases
* Patients whose permanent central incisor and permanent first molar teeth had not erupted

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 202 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
Simplified Oral Hygiene Index (OHI-S) Scoring | 30 days
  In the present study, 30 days after verbal and video-based oral hygiene instructions were given to patients, oral hygiene status was similarly determined and recorded using OHI-S index method (OHI-S final scores).

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Demirel A, Guclu HS, Guclu M, Bagis N. Evaluation of Effects of Verbal and Video-Based Instructions on the Improvement of Oral Hygiene Status in Children: A Randomised Clinical Trial. Int J Dent Hyg. 2025 Aug;23(3):575-583. doi: 10.1111/idh.12898. Epub 2025 Jan 29. PMID 39887898